CLINICAL TRIAL: NCT06720584
Title: WHEEL: Improving Quality of Life in SLE by Stratified Personalized Health Planning
Brief Title: Whole Health Empowerment for Endotypes of Lupus: Improving Quality of Life in SLE
Acronym: WHEEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00111699; W81XWH-22-1-0611 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-11-12; First posted 2024-12-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: systemic lupus erythematosus; SLE; Type 2 SLE; health coach; support program; mindfulness; fatigue; brain fog; pain
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Fatigue; Mental Fatigue; Pain

STUDY DESIGN:
Intervention Model Description: Pilot randomized wait-list controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Immediate Treatment (Experimental): Group 1 participants receive the intervention first which is completing the 4-month program. They will receive an additional survey when Group 2 completes the intervention.
  Interventions: Behavioral: Health coach-led, online support program for people living with lupus
- Group 2: Wait-List Control (Delayed Intervention) (Other): Group 2: Wait-List Control (Delayed Intervention) does not get the intervention while Group 1 is getting the intervention. Group 2 receives the intervention AFTER Group 1 has completed the intervention.
  Interventions: Behavioral: Health coach-led, online support program for people living with lupus

INTERVENTIONS:
Behavioral: Health coach-led, online support program for people living with lupus — The health coach-led online support and education program for people living with lupus. It includes 8 group sessions and 2 individual sessions with the health coach to set individual goals. Each program group will include up to 10 participants.
  Program Session Structure (~60-75 minutes): educational component presented using a slide set, discussion questions interspersed, mindfulness activities, goal check-ins.
  Associated Materials: Notebook, expert videos available.

SUMMARY:
For people living with people living with systemic lupus erythematosus (SLE) the symptoms with the largest impact on their quality of life - fatigue, pain, and brain fog - are not always addressed in rheumatology clinic visits. To address the quality-of-life limitations, the investigators have created and will test the health coach-led, 8-session Whole Health Empowerment for Endotypes of Lupus (WHEEL) online support program. This program moves beyond traditional clinic visits and standard educational curricula to engage patients in creating their own health goals and therapeutic plans in a setting that emphasizes both the psychosocial and clinical factors contributing to disease. Participants will attend the virtual sessions, work with their health coach on two additional sessions, and complete surveys.

DETAILED DESCRIPTION:
The investigators have created the WHEEL Program* (explained below) based on a previously developed Personalized Health Planning model, patient surveys, patient and provider focus groups feedback for WHEEL curricula and materials, and a User Testing of the WHEEL Program. The objective is to assess the feasibility of the WHEEL program, including its acceptability, demand, implementation, practicality, integration, and preliminary efficacy as an approach to improve quality of life in people with SLE. Our working hypothesis is that the WHEEL protocol will be feasible and acceptable to patients with SLE and demonstrate initial efficacy for improving quality of life. The investigators expect, however, that patients with Intermittent and Persistent Type 2 SLE* (see description below) will experience improvement in different domains of quality of life based on their initial deficits and the content of each program. At the completion of this proposal, the investigators will have a tested, feasible, and expandable protocol that the investigators will be prepared to test in larger SLE populations. This work represents a dramatic breakthrough for SLE self-management programs, tailoring the program to the specific SLE endotypes, providing essential group support, and empower patients with SLE to take control of their disease to improve their quality of life.

WHEEL Program Key Elements:

1. Eight, virtual, bi-weekly group sessions, ~ 60-90 minutes per session
2. Program facilitated by a certified health coach with clinical licensure and supported by a co-facilitator
3. Themed group sessions focusing on understanding disease, medications and symptoms, motion/exercise, sleep/rest, nutrition, mindfulness/stress management, and personal goals.
4. Curriculum comprised into a patient notebook with interactive and educational content, activities, and figures that mirror the information and activities that comprise the group sessions.
5. Each group session includes interactive activities, health coaching, goal progress tracking, mindfulness-based practices, group discussion, social support, and empathy and empowerment between patients
6. One-on-one consultation with health coach to develop a Personal Health Plan supported by shared patient-provider health assessments (i.e., Patient Health Self-Assessment and Provider Health Risk Assessment)
7. Follow-up one-on-one consultation with the health coach to enhance engagement through motivational coaching based on patient-identified priorities and health goals.

Description of Type 1 and 2 SLE symptoms, Intermittent and Persistent Type 2 SLE:

A team of clinicians and investigators within the Duke Lupus Clinic developed a new approach to SLE care by creating the Type 1 & 2 SLE Model. In this model, signs and symptoms of SLE are divided into two broad categories. Type 1 SLE symptoms consist of what is classically considered SLE activity and recorded in provider-reported measures of SLE activity, including synovitis, cutaneous lupus, nephritis, and other objective signs. Type 2 SLE symptoms include fatigue, myalgia, mood disturbance, and cognitive dysfunction. Duke researchers further refined the model and propose two endotypes of SLE: Intermittent Type 2 SLE (correlation between Type 1 & 2 SLE symptoms, with both sets of symptoms worsening and improving around the same time) and Persistent Type 2 SLE (omnipresent Type 2 SLE symptoms that do not fluctuate when they have flares of Type 1 SLE).

ELIGIBILITY:
Inclusion Criteria.

(1) enrolled in the Duke Lupus Registry* for ≥1 year; (2) had ≥ 3 visits in the Duke Lupus Registry, (3) attended a Duke Lupus clinic visit in the last year, (4) meets Type 1 & 2 SLE Activity criteria as defined below, (5) meets Persistent Type 2 SLE or Intermittent Type 2 SLE criteria as described below, (meets classification criteria for SLE (SLICC, ACR, or EULAR/ACR)), (7) female.

* Active Type 1: SLEDAI ≥6, clinical SLEDAI ≥4, Type 1 PGA ≥1, or active lupus nephritis
* Active Type 2: PSD: ≥8 or Type 2 PGA ≥1
* Persistent Type 2 SLE: Active Type 2 SLE at 3 visits, Active Type 1 SLE at 0-2 visits
* Intermittent Type 2 SLE: Active Type 2 SLE at 1-2 with Active Type 1 SLE at 1-3 visits

Participants will be stratified based on their Type 2 SLE activity in the prior 3 Duke Lupus Clinic visits as defined above.

* Duke Lupus Registry participants must be age ≥18 years; disease duration of ≥1 year; ability to speak and read English; able to consent themselves

Exclusion Criteria:

(1) significant cognitive impairment as determined by the treating rheumatologist; (2) untreated serious mental illness; (3) inability to provide informed consent; (4) participation in Aim 2 WHEEL curriculum development; (5) does not commit to attending sessions and using a tablet/computer. All participants will provide e-consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Participant Satisfaction | Post-intervention (within four weeks of intervention ending)
  o Study-specific survey asking participants about their satisfaction on a scale from 0=completely unsatisfied to 10=completely satisfied
Intervention Adherence | 10-months post-baseline
  Total number of group sessions and health coach sessions attended.
Survey Completion | 10-months post-baseline
  Count the total number of surveys completed at 10 months post-baseline. Participants are to complete 2 surveys, LupusPRO and Whole Health Assessments pre-intervention, and 2 surveys, LupusPRO and Whole Health Assessments post-intervention.
  The range of completed surveys is 0-4 surveys, 0-100% complete. Completion of the entire survey is counted as completed.

SECONDARY OUTCOMES:
Participant Accrual | Baseline
  Number of participants consented to the study.
Participant Attrition | 10-months post-baseline
  Number of consented participants who withdrew/were withdrawn from the program.

OTHER OUTCOMES:
Change in LupusPro | Baseline, 5-months post baseline, and 10-month post-baseline
  LupusPro is a 43-question quality of life survey designed specifically for patients with lupus. It measures ways that lupus may affect a patient's mental, emotional and physical health. Scores range from 0 -100 and higher scores indicate higher quality of life.
Change in Whole Health Assessment | Baseline, 5-months post baseline, and 10-month post-baseline
  Whole Health Assessment assesses 10 components of everyday life that can affect their overall health. Scores range from 0 -100 and higher scores indicate areas of strength.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rogers, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT06720584/ICF_000.pdf